CLINICAL TRIAL: NCT02760836
Title: Development and Validation of Predictive Model of Clinical Outcomes Using Pattern Analysis of Web-based Self-reporting Symptom Diary for Crohn's Disease
Brief Title: Predictive Model of Clinical Outcomes Using Web-based Self-reporting Symptom Diary for Crohn's Disease
Acronym: PICASSO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Kyungpook National University Hospital (Other)
Responsible Party: Principal Investigator, Eun Soo Kim, MD, PhD, Professor, Kyungpook National University Hospital
Other Study IDs: KNUH2016-03-030
Record Dates: First submitted 2016-05-02; First posted 2016-05-04 (Estimated); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: Crohn's Disease
Keywords: Crohn's disease; disease outcomes
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to develop and validate a predictive model of clinical outcomes based on the results of web-based self-reporting symptom diary for Crohn's disease.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed of Crohn's disease within 6 months
* Must record their symptom in a web-based symptom diary at least 4 consecutive times for 2 months.

Exclusion Criteria:

* Not able to use smart phone.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Crohn's disease from 4 tertiary referral centers.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2016-04 (Actual); Primary Completion 2020-04 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Hospitalization | 2 years
Unscheduled visit | 2 years

SECONDARY OUTCOMES:
Bowel resection surgery | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Eun Soo Kim, MD, PhD, Principal Investigator — Kyungpook National University Hospital
Locations (1):
- Kyungpook National University Hospital, Daegu, South Korea

IPD SHARING:
Plan to Share IPD: No